CLINICAL TRIAL: NCT00148759
Title: A Switch From Twice Daily to Once Daily Lopinavir/Ritonavir: A 24-hour Pharmacokinetic Profile to Evaluate Sex Differences
Brief Title: Kaletra Sex/Gender Pharmacokinetics (PK) Study
Acronym: LPVGenderPK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Ighovwerha Ofotokun, Associate Professor of Medicine, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002448; UPN 04092824 (Other Grant/Funding Number: Abbott Virology); GCRC0605G (Other: Other)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Sex differences; Pharmacokinetic; Lopinavir/ritonavir; Treatment Experienced; HIV-infection
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- adult male subjects (Active Comparator): LPV/r 800/200 mg once daily
  Interventions: Drug: LPV/r
- Adult female subjects (Experimental): LPV/r 800/200 mg once daily
  Interventions: Drug: LPV/r

INTERVENTIONS:
Drug: LPV/r — LPV/r 800/200 mg once daily
  Other Names: Daily LPV/r; Kaletra

SUMMARY:
The levels of lopinavir achieved in the blood following oral ingestion of standard doses of Kaletra (lopinavir/ritonavir) in HIV-infected men was compared with those achieved in HIV-infected women receiving the same dose of the drug.

DETAILED DESCRIPTION:
The association between patient sex and the tolerability of antiretroviral drugs (ARVs) is increasingly being recognized. Several lines of evidence suggest that women are more likely than men to develop side effects to ARVs. On the other hand, it has been generally accepted that the efficacies of the ARVs are similar in both sexes. However, recent studies suggest that this may not always be the case. In addition to these observed sex-related differences in the effects of ARVs, there is growing evidence that the pharmacokinetic profile of some of these drugs may be different among male and female HIV infected patients.

The fact that female sex is a risk factor for enhanced antiretroviral effects (including toxicities) has an important implication, particularly from a global health perspective as women now represent the fastest growing segment of the HIV/AIDS epidemic. Therefore, an understanding of the magnitude, clinical significance, and the mechanisms underlying this phenomenon deserves further study. Knowledge acquired from such studies will likely contribute to improved survival among female HIV-infected patients, through optimization of antiretroviral therapeutic regimens in manners that minimize serious adverse effects and improve adherence.

Similarly, the influence of race on the pharmacological effects of ARVs deserves further investigation. Although, there is no reason to believe based on available evidence that racial differences exist in the pharmacological effects of ARVs, the need however exists to explore the influence of race on ARVs pharmacokinetics and treatment outcomes. This is so because data on race related differences on ARV effects is limited, and in addition, people of ethnic minority have been disproportionately under represented in clinical trials involving these drugs in spite of the fact that they bear a larger burden of the HIV epidemic.

Our study will examine the influence of race and sex on the 24-hr pharmacokinetics of lopinavir/ritonavir (an antiretroviral agent commonly used in naïve patients) following a switch from LPV/r 400/100 mg twice daily to 800/200 mg once daily dosing. Tolerability (measured by toxicity grade of diarrhea) and change in quality of life following switch from twice daily to once daily dosing will also be assessed using appropriate validated measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years
* Diagnosis of HIV infection as previously established by HIV Enzyme-Linked Immunosorbent Assay (ELISA) test and confirmed by Western blot analysis.
* Must have been taking LPV/r as part of an antiretroviral regimen at a dose of 400/100 mg orally twice per day for at least 3 months.
* Recent (within last 90 days) HIV-RNA copies must be less than 400 copies/ml

Exclusion Criteria:

* Hepatic abnormality: alanine-aminotransferase (ALT), aspartate-aminotransferase (AST) or total bilirubin (TBR) ≥ 3 x upper limit of normal
* Renal insufficiency: serum creatinine ≥ 2 mg/dl
* Co-infection with hepatitis B and/or C viruses
* Pregnant or breastfeeding
* Use of concurrent medications known to affect lopinavir or ritonavir concentrations significantly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igho Ofotokun, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Program, Atlanta, Georgia, United States

REFERENCES:
- [Result] Ofotokun I, Chuck SK, Binongo JN, Palau M, Lennox JL, Acosta EP. Lopinavir/Ritonavir pharmacokinetic profile: impact of sex and other covariates following a change from twice-daily to once-daily therapy. J Clin Pharmacol. 2007 Aug;47(8):970-7. doi: 10.1177/0091270007302564. Epub 2007 Jul 5. PMID 17615254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Grady Infectious Diseases Clinic in Atlanta, Georgia between June 2005 and January 2007. All subjects provided written informed consent before undergoing any study procedures.
Pre-assignment Details: Of the 23 subjects enrolled, 20 completed the study including the PK sampling. Three subjects (2 males and 1 female) dropped out. Two subjects were unavailable for the 24-hour PK sampling because of changes in their work schedules, and the third subject was lost to follow-up after the initial study visit.
Groups:
- Male Arm: Male subjects
- Female Arm: Female subjects
Period: Overall Study
Arm/Group | Male Arm | Female Arm
Started | 11 | 12
24-hr PK Sampling | 9 | 11
Completed | 9 | 11
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Male subjects
- Group 2: Female subjects
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (16) | 39 (18) | 38 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 12
  Male | 11 | 0 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Secondary Outcome: 24-hr LPV Cmax
Description: LPV Cmax at Steady State
Time Frame: 24 hours
Measure: Geometric Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 11
ng/mL | 12417 [11622 to 13699] | 12271 [7219 to 14113]

2. Primary Outcome: 24-hr LPV AUC
Description: Steady state(2 weeks after therapy change)
Time Frame: 24 hours
Measure: Geometric Mean (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 11
ng*hr/mL | 142,160 [136300 to 191390] | 152140 [110840 to 214180]

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes